CLINICAL TRIAL: NCT00887042
Title: Phase II Study of Reduced Toxicity Myeloablative Conditioning Regimen for Cord Blood Transplantation in Pediatric Acute Myeloid Leukemia
Brief Title: Study of Reduced Toxicity Myeloablative Conditioning Regimen for Cord Blood Transplantation in Pediatric AML
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Korean Society of Pediatric Hematology Oncology (Network)
Responsible Party: The Korean Society of Hematology, The Korean Society of Pediatric Hematology Oncology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSPHO-S0501
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Cord blood transplantation; Pediatric
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; Busulfan; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fludarabine (Experimental)
  Interventions: Drug: Fludarabine, Busulfan, Thymoglobulin

INTERVENTIONS:
Drug: Fludarabine, Busulfan, Thymoglobulin — fludarabine (40 mg/m2 once daily i.v. on days -8, -7, -6, -5, -4 & -3) busulfan (0.8 mg/kg every 6 hours i.v. on days -6, -5, -4, & -3) thymoglobulin (2.5 mg/kg once daily i.v. on days -8, -7, & -6)

SUMMARY:
Cord blood transplantation (CBT) is an alternative option for patients with pediatric acute leukemia that indicated stem cell transplantation. Although CBT is as affective as unrelated bone marrow transplantation with lower graft versus host disease (GVHD) severity and incidence, transplantation related mortality (TRM) has been major problems after myeloablative conditioning. To reduce TRM, CBT with non-myeloablative conditionings have been performed but not so satisfactory especially for engraftment rate. Recently reduced toxicity myeloablative conditioning regimen was developed with promising result in adult bone marrow or mobilized peripheral blood transplantation. To increase the engraftment potential with low TRM rate, reduced toxicity myeloablative conditioning composed of fludarabine, intravenous busulfan plus thymoglobulin is planned for pediatric patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
Since the first successful transplantation using umbilical cord blood (UCB) to treat a patient with Fanconi anemia in 1988 (Gluckman E, 1989), cord blood transplantation (CBT) has become an alternative to bone marrow transplantation (BMT) to treat a variety of diseases. Cord blood cells have many theoretical advantages as grafts for stem cell transplantation because of the immaturity of newborn cells. Compared to adults, UCB stem cells produce larger in vitro hematopoietic colonies, are able to expand in long-term culture in vitro (Ahn HS, 2003). The properties of UCB cells should theoretically compensate for the relatively low number of cells obtained in a single UCB unit and, through rapid expansion, reconstitute myeloablated patients with fewer nucleated cells (by 1-2 logs) than bone marrow (Barker JN, 2003-1).

Recent results of CBT revealed that HLA-matched and 1-antigen mismatched unrelated CBT had similar survival as HLA-matched unrelated BMT and both the cell dose and HLA-disparity influenced the outcome of CBT (CIBMTR data). But the major problems of CBT were engraftment failure and transplantation related mortality (TRM) that compromised the outcomes of CBT. As the numbers of stem cells are lower and immune cells are immature in cord blood than bone marrow, the engraftment and immunologic recovery are delayed in CBT than BMT and these properties of CBT result in higher rate of TRM up to 39% during 100 days after CBT (Rocha V, 2001). Early results of CBT also reported upto 50% of TRM (Gluckman E, 1997; Rubinstein P, 1998) and CIBMTR also reported that the cumulative incidence of TRM in pediatric study is about 40%.

As the TRM is higher in CBT especially after conventional myeloablative conditioning, non-myeloablative conditioning regimens are investigated especially for adult CBT (Barker JN, 2003-2; Chao NJ, 2004). But studies about pediatric acute leukemia patients are not so much and our pilot data suggested that CBT with non-myeloablative conditioning resulted in lower engraftment rate and anti-leukemic effect although with low morbidity and mortality (Ahn HS, 2004).

Recently, fludarabine based reduced toxicity myeloablative regimens were investigated with promising result in adult transplant with bone marrow or mobilized peripheral blood (Russell JA, 2002; Bornhauser M, 2003; de Lima M, 2004).

Purine-analog, in particular fludarabine, has some advantage over cyclophosphamide. It has immunosuppressive property that allows the engraftment of hematopoietic stem cells with minimal extramudullary toxicity. Fludarabine also inhibit the repair mechanism of alkylating agent induced DNA damage, thus providing a synergistic effect if pre-exposed to the target tissue.

As the fludarabine plus myeloablative dose of busulfan allowed good engraftment and reduced toxicity in transplant with bone marrow or mobilized peripheral blood, this combination could be optimal for the conditioning regimen for CBT, which has high TRM and lower engraftment rate with conventional myeloablative conditioning.

To increase the engraftment potential with low TRM rate, reduced toxicity myeloablative conditioning composed of fludarabine, intravenous busulfan, thymoglobulin for CBT is planned for pediatric patients with AML.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute myeloid leukemia (FAB or WHO classification).
2. Indicated for hematopoietic stem cell transplantation.
3. Age: < 21 years old.
4. Performance status: ECOG 0-2.
5. Patients must be free of significant functional deficits in major organs, but the following eligibility criteria may be modified in individual cases. 1. Heart: a shortening fraction > 30%, ejection fraction > 45%. 2. Liver: total bilirubin < 2 × upper limit of normal; ALT < 3 × upper limit of normal. 3. Kidney: creatinine <2 × normal or a creatinine clearance (GFR) > 60 ml/min/1.73m2.
6. Patients must lack any active viral infections or active fungal infection.
7. Appropriate cord blood unit is available: accept HLA mismatch in two of six loci (pairs of A, B, and DR). Allow 2 units cord transplantation.
8. One of parents should sign informed consent.

Exclusion Criteria:

1. Pregnant or nursing women.
2. Malignant (except acute myeloid leukemia) or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
3. Psychiatric disorder that would preclude compliance.
4. More than three HLA type mismatch.
5. T cell depleted or ex vivo expanded cord blood.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2006-06; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate the engraftment potential of fludarabine, busulfan plus thymoglobulin conditioning regimen for CBT in AML. | From June 2006 to May 2010
To evaluate the incidence and severity of toxicity and treatment related mortality. | From June 2006 to May 2010

SECONDARY OUTCOMES:
To evaluate overall and event free survival rate. | From June 2006 to May 2010
To evaluate acute and chronic GVHD. | From June 2006 to May 2010
To evaluate immunologic recovery after CBT. | From June 2006 to May 2010

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Seop Ahn, M.D, Ph. D, Principal Investigator — The Korean Society of Pediatric Hematology Oncology
Locations (1):
- Seoul National University Hospital, Seoul, Chongno-gu, South Korea